CLINICAL TRIAL: NCT05564429
Title: Assessment of [18F]SF12051 for Imaging the 18-kDa Translocator Protein (TSPO) in Brain and Whole Body of Healthy Subjects
Brief Title: [18F]SF12051 for Imaging the 18-kDa Translocator Protein (TSPO) in Brain and Whole Body of Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to futility
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000674; 000674-M
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: PET Imaging; Neuroinflammation; Tspo
MeSH Terms: conditions — Neuroinflammatory Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High affinity binder (HAB) Translocator Protein (TSPO) genotype (Experimental): Healthy participants with HAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body or brain positron emission tomography (PET) scan. Participants were randomized to either phase 1, 2, or 3. Phases 1 & 3 had whole body PET scan and phase 2 had brain PET scan.
  Interventions: Drug: 18F-SF12051
- Low affinity binder (LAB) Translocator Protein (TSPO) genotype (Experimental): Healthy participants with LAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body or brain positron emission tomography (PET) scan. Participants were randomized to either phase 1, 2, or 3. Phases 1 & 3 had whole body PET scan and phase 2 had brain PET scan.
  Interventions: Drug: 18F-SF12051
- Mixed affinity binder (MAB) Translocator Protein (TSPO) genotype (Experimental): Healthy participants with MAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body or brain positron emission tomography (PET) scan. Participants were randomized to either phase 1, 2, or 3. Phases 1 & 3 had whole body PET scan and phase 2 had brain PET scan.
  Interventions: Drug: 18F-SF12051

INTERVENTIONS:
Drug: 18F-SF12051 — Injected intravenously followed by PET scanning

SUMMARY:
Background:

Inflammation in the brain plays a role in many diseases. Being able to measure inflammation in a person's brain might help to diagnose and treat these diseases. One protein (TSPO) appears in higher numbers when inflammation affects the brain. To see TSPO when a person's body is scanned, researchers need a substance called a radiotracer that will attach to this protein and no other molecules.

Objective:

This study will test whether a new radiotracer ([18F]SF12051) can make TSPO appear on PET scans of a person's brain and body.

Eligibility:

Healthy people aged 18 and older.

Design:

This study requires 2 to 4 visits to the clinic.

All participants will be screened. They will have a physical exam. They will have blood tests and a test of their heart function.

Some participants will have a positron emission tomography (PET) scan of the whole body. The radiotracer will be injected through a tube (catheter) placed in a vein in the arm. The PET scanner is a machine shaped like a doughnut. Participants will lie on a bed that slides in and out of the scanner. The scan will take about 2 hours.

Some participants will have a PET scan of just their head. After they are injected with the radiotracer, they will lie on a bed with their head in the scanner. Blood will be drawn from a catheter in the wrist during the scan.

Some participants will have a magnetic resonance imaging (MRI) scan of the brain. They will lie on a narrow bed that slides into a tube.

DETAILED DESCRIPTION:
Study Description:

This study is intended to provide information on the novel [18F]SF12051 radioligand and its ability to localize and measure TSPO in the brain and body of healthy individuals.

Objectives:

Primary Objective: To study the brain uptake of [18F]SF12051 and perform kinetic modeling of the [18F]SF12051 in the three different TSPO genotypes.

Secondary Objectives: To study the brain retest characteristics, biodistribution and dosimetry of [18F]SF12051 in healthy subjects.

Endpoints:

Primary Endpoint: The distribution volume of the radioligand and stability over time calculated with compartmental modeling, attention paid to differences in mean distribution volumes between TSPO genotypes for determining genotype sensitivity.

Secondary Endpoints: Retest variability and reliability and organ time- activity curves to determine biodistribution and dosimetry.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged 18 years or older.
* Healthy based on medical history, physical examination, and laboratory testing.
* Able to provide informed consent.
* Willing and able to complete all study procedures.
* Have been screened for TSPO genotype under 01-M-0254 "The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Participants".
* Have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists*.
* Agree to adhere to the lifestyle considerations

  * Does not apply to Phase 1 and 3 participants as they will not have an arterial line.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Clinically significant abnormalities on EKG or laboratory testing. This includes CBC; acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen); hepatic panel (alkaline phosphatase, ALT, AST, bilirubin total, and bilirubin direct); mineral panel (albumin, calcium, magnesium, phosphorus); prothrombin and partial prothrombin tests.
* Participants should not have taken NSAIDs or willow bark tea for two weeks prior to the PET scan.
* Any current Axis I diagnosis.
* Positive test for HIV.
* Unable to have an MRI scan*.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* History of seizures, other than in childhood and related to fever.
* Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours, including claustrophobia and weight greater than the maximum for the scanner (500 lbs).
* Pregnancy or breast feeding.
* Able to get pregnant but does not use birth control.
* Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use affects the function of daily life.
* Unable to travel to NIH.
* National Institute of Mental Health (NIMH) staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

  * Phase 1 and 3 participants will not get an MRI.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.The results will be submitted to ClinicalTrials.gov
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol
Access Criteria: BTRIS

REFERENCES:
- [Derived] Yan X, Simeon FG, Liow JS, Morse CL, Jana S, Montero Santamaria JA, Jenkins M, Zoghbi SS, Pike VW, Innis RB, Zanotti-Fregonara P. [18F]SF51, a novel 18F-labeled PET radioligand for translocator protein 18kDa (TSPO) in brain, works well in monkeys but fails in humans. J Cereb Blood Flow Metab. 2025 Feb;45(2):365-372. doi: 10.1177/0271678X241304924. Epub 2024 Dec 9. PMID 39654356
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000674-M.html

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Started | 0 | 0 | 1
Whole Body PET Scan | 0 | 0 | 1
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Started | 3 | 2 | 3
Brain PET Scan | 3 | 2 | 3
Completed | 3 | 2 | 3
Not Completed | 0 | 0 | 0
Period: Phase 3
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Started | 1 | 0 | 0
Whole Body PET Scan | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype: Healthy participants with HAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body or brain positron emission tomography (PET) scan.
- Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype: Healthy participants with LAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body or brain positron emission tomography (PET) scan.
- Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype: Healthy participants with MAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body or brain positron emission tomography (PET) scan.
- Total: Total of all reporting groups
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype | Total
Number analyzed (Participants) | 4 | 2 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 4 | 10
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 3 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 2 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 3 | 7
  White | 0 | 2 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Whole Body PET Uptake of [18F]SF12051 - Phase 1
Description: Participant received whole body PET scan and Uptake of [18F]SF12051 was measured using the Siemens Biograph mCT. Organ dosimetry was measured as microsieverts per mega-becquerel (uSv/MBq).
Time Frame: Up to 120 minutes during the scan
Population: Participant who completed phase 1 of the study. Whole body PET imaging was done for one subject with a low injection activity of ~2 mCi to confirm that no organ has prominently high uptake of [18F]SF12051.
Measure: Number; unit: uSv/MBq
Groups:
- Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype: Healthy participants with MAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body PET scan.
Arm/Group | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Number analyzed (Participants) | 1
uSv/MBq
  Brain | 6
  Heart | 17
  Liver | 8
  Kidneys | 16
  Lungs | 11
  Stomach | 18
  Spleen | 15
  Bone Marrow | 15
  Gallbladder | 16
  Small intestine | 25
  Testicles | 14
  Urinary bladder | 21
  Whole body | 15

2. Primary Outcome: Brain PET Uptake of [18F]SF12051 - Phase 2
Description: Participant received brain PET scan and Uptake of [18F]SF12051 was measured using the Siemens Biograph mCT. Volume of distribution (Vt) was calculated via 2-Tissue-Compartment Model with plasma input function.
Time Frame: Up to 120 minutes during the scan
Population: All participants who completed phase 2 of the study. Data for one participant was not useable.
Measure: Mean (Standard Deviation); unit: mL*cm-3
Groups:
- High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype: Healthy participants with HAB TSPO genotype receive 18F-SF12051 intravenously followed by brain positron emission tomography (PET) scan.
- Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype: Healthy participants with LAB TSPO genotype receive 18F-SF12051 intravenously followed by brain positron emission tomography (PET) scan.
- Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype: Healthy participants with MAB TSPO genotype receive 18F-SF12051 intravenously followed by brain positron emission tomography (PET) scan.
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Number analyzed (Participants) | 3 | 2 | 2
mL*cm-3 | 0.833333333 (0.328) | 0.40 (0.0225) | 0.90 (0.036)

3. Primary Outcome: Whole Body PET Uptake of [18F]SF12051 - Phase 3
Description: as for outcome 1
Time Frame: Up to 120 minutes during the scan
Population: Participant who completed phase 3 of the study.
Measure: Number; unit: uSv/MBq
Groups:
- High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype: Healthy participants with HAB TSPO genotype receive 18F-SF12051 intravenously followed by whole body PET scan.
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype
Number analyzed (Participants) | 1
uSv/MBq
  Brain | 5
  Heart | 15
  Liver | 12
  Kidneys | 17
  Lungs | 13
  Stomach | 15
  Spleen | 10
  Bone Marrow | 12
  Gallbladder | 20
  Small intestine | 20
  Ovaries | 15
  Urinary bladder | 12
  Whole body | 15

4. Secondary Outcome: Area Under the Organ Time-Activity Curves From 0-120 - Phase 1
Description: Biodistribution and dosimetry of [18F]SF12051 in healthy subjects was measured as area under the curve from 0-120 minutes shown as concentration of radioactivity reported as standard uptake values (SUV) x time during the course of the scans for each organ.
Time Frame: Up to 120 minutes during the scan
Population: Participant who completed phase 1 of the study.
Measure: Number; unit: SUV*minutes
Arm/Group | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Number analyzed (Participants) | 1
SUV*minutes
  Brain | 84.78437744
  Heart | 497.9329916
  Liver | 357.8754055
  Kidneys | 345.5662222
  Lungs | 93.28630134
  Stomach | 348.3474892
  Spleen | 438.5340085
  Urinary bladder | 271.9311702
  Bone Marrow | 868.883177
  Gallbladder | 152.5233703
  Small intestine | 218.0137982
  Testicles | 71.86889245

5. Secondary Outcome: Area Under the Organ Time-Activity Curves From 0-120 - Phase 3
Description: as for outcome 4
Time Frame: Up to 120 minutes during the scan
Population: Participant who completed phase 3 of the study
Measure: Number; unit: SUV*minutes
Arm/Group | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Number analyzed (Participants) | 1
SUV*minutes
  Brain | 56.6832231
  Heart | 491.710075
  Liver | 141.3314325
  Kidneys | 215.9146934
  Lungs | 92.14993947
  Stomach | 170.0881894
  Spleen | 238.9553087
  Urinary bladder | 234.1664917
  Bone Marrow | 230.539214
  Gallbladder | 115.1009919
  Small intestine | 144.9270488
  Ovaries | 67.67155656

6. Secondary Outcome: Test-Retest Variability of [18F]SF12051
Description: Assess test-retest variability of [18F]SF12051 using absolute test-retest variability (aTRV).
  aTRV = | retest value - test value| / (test value + retest value) * 200%
Time Frame: Up to 120 minutes during the scan
Population: Data were not collected due to termination of the study
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Test-Retest Reliability of [18F]SF12051
Description: Assess test-retest reliability of [18F]SF12051 using intraclass correlation coefficient (ICC)
  ICC = (between-subject standard deviation)^2/[(between-subject standard deviation)^2 + (within-subject standard deviation)^2]
Time Frame: Up to 120 minutes during the scan
Population: Data were not collected due to termination of the study
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to five day post PET scan visit
Arm/Group | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Affinity Binder (HAB) Translocator Protein (TSPO) Genotype (N=4) | Low Affinity Binder (LAB) Translocator Protein (TSPO) Genotype (N=2) | Mixed Affinity Binder (MAB) Translocator Protein (TSPO) Genotype (N=4)
Pain (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT05564429/Prot_SAP_000.pdf